CLINICAL TRIAL: NCT04944940
Title: An Observational Study to Assess Clinical, Molecular and Imaging Biomarkers in Spinal and Bulbar Muscular Atrophy (SBMA)
Brief Title: Clinical, Molecular and Imaging Biomarkers in Spinal and Bulbar Muscular Atrophy (SBMA)
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000428; 000428-N
Record Dates: First submitted 2021-06-29; First posted 2021-06-30 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06-30

CONDITIONS: Spinal and Bulbar Muscular Atrophy; Kennedys Disease; Motor Neuron Disease
Keywords: Motor Neuron Disease; Spinal and Bulbar Muscular Atrophy; Kennedys disease; Androgen Receptor; Natural History Study; Natural History
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy male participants who are age and sex matched to the SBMA participants
- Patients with Spinal and bulbar muscular atrophy (SBMA): Male participants with genetically confirmed SBMA

SUMMARY:
Background:

SBMA is an inherited chronic disease. It affects males in mid to late adulthood. It causes slowly progressive weakness of muscles and hand tremors. Researchers want to learn more about the effects of SBMA.

Objective:

To identify measurements that change over time in SBMA, including tests of muscle strength and function, as well as measurements of muscle and fat size.

Eligibility:

Men over the age of 18 both with and without a history of SBMA.

Design:

Participants will have a medical history, physical exam, and blood and urine tests. They will have neuromuscular ultrasound. They will have a lumbar puncture to obtain spinal fluid. For this, a needle will be inserted into the spinal canal in the lower back.

Participants will have muscle strength and function tests. These tests may include pushing, pulling, rising from a chair and sitting back down, and/or walking. During these tests, they may wear an accelerometer (activity tracker) on their wrist.

Participants will get an activity tracker to wear on their wrist for 10 days at home every 3 months.

Participants with SBMA will also have lower limb magnetic resonance imaging (MRI) and optional whole-body MRI. They will have lung function tests. They will have speech and swallow tests. They will complete questionnaires. They may have optional body scans to measure bone density and lean body mass. They may have optional muscle biopsies. For biopsies, a needle will be used to take a small piece of muscle from the leg.

Participants with SBMA will have 5 study visits over 2 years (every 6 months). Participants without SBMA will have 1 study visit.

DETAILED DESCRIPTION:
Study Description:

Spinal and bulbar muscular atrophy (SBMA) is an inherited form of motor neuron disease caused by a CAG-repeat expansion in the androgen receptor gene on the X chromosome for which there is no treatment currently. Biomarkers will be collected from participants with SBMA during this study to understand the natural history and progression of the disease.

Objectives:

The main objective of this study is to develop clinical, molecular and imaging outcome parameters that correlate with disease progression and severity and that predict clinical decline. These biomarkers and outcome measures can serve as potential tools for the evaluation of efficacy in future therapeutic studies in SBMA.

Endpoints:

The studies performed under this protocol are exploratory. However, the following measures may be used to characterize baseline status and disease progression over the course of the study:

Muscle strength by manual and quantitative myometry

Distance traveled in meters on the 6-minute walk test

Activity levels and parameters of gait as measured by accelerometers

Global disability measured by the SBMAFRS questionnaire and other tools/instruments

Fatigue as measured by the Fatigue Severity Scale

Breathing function measured by pulmonary function test

Swallow and speech function measured by questionnaires, tongue muscle strength, digital audio recordings for analysis of voice and speech, and barium swallow

Skeletal muscle MRI measurement of muscle volume and fat fraction

Whole body MRI measurement of body muscle fat fraction, muscle fat infiltration, and liver.

Skeletal muscle ultrasound measurement of muscle thickness, echogenicity and elasticity

Nerve ultrasound measurement of nerve cross sectional area and anterior posterior diameter

Laboratory studies from blood, serum, urine, stool, and CSF

Muscle biopsy assessment of androgen receptor levels and function

ELIGIBILITY:
* INCLUSION CRITERIA:

Some restrictions are placed on participation in the study because we aim to identify disease biomarkers specific to those with early to intermediate stages of disease who would be potential candidates for future therapeutic studies.

In order to be eligible to participate in the SBMA cohort, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male, above the age of 18 years
* Genetically confirmed SBMA
* Ability of subject to understand and the willingness to sign a written informed consent document
* Ability of subject to travel to the NIH Clinical Center.

Note: an SBMA patient who meets both of the additional following criteria will be offered an optional whole body MRI at subsequent follow-up visits:

* Spinal bulbar muscular atrophy functional rating of < 50 (and > 35).
* On initial whole body MRI, subject has evidence of muscle fat replacement such that the total volume of disease affected muscles (i.e., muscles with at least 10% muscle fat infiltration and no more than 50% muscle fat fraction) is at least:

  * 500ml if only 1 muscle is eligible or
  * 250ml if more than one muscle meets the criteria

In order to be eligible to participate in this study in the Healthy Control cohort, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures and availability to travel to the NIH for the duration of the study
* Male, above the age of 18 years
* No history of SBMA or other neuromuscular disorder
* No history of facial palsy
* Ability of subject to understand and the willingness to sign a written informed consent document
* Ability of subject to travel to the NIH Clinical Center.

EXCLUSION CRITERIA:

SBMA is a disease that affects males and manifests in adulthood. Thus, woman and children are not included in this study. This study will not include individuals who lack consent capacity.

An SBMA patient who meets any of the following criteria will be excluded from participation in this study:

* Contraindications to MRI such as a contraindicated non-removable metal device (i.e., pacemaker, defibrillator, insulin pump, metal clips, non-removable jewelry) or claustrophobia.
* Non ambulatory
* Use of androgen reducing agents within the past two years

Note: An SBMA patient who meets any of the following criteria will be excluded from the lumbar puncture procedure:

* PT/PTT values that are prolonged greater than or equal to 3 seconds from the upper limit of normal (including treatment with oral and parenteral anticoagulants)
* INR greater than or equal to 1.5, thrombocytopenia (<70,000), or abnormal bleeding time or platelet dysfunction
* History of a bleeding disorder
* Use of anticoagulants

Note: An SBMA patient who meets any of the following criteria will be excluded from the muscle biopsy procedure:

* Advanced wasting of tibialis anterior that precludes needle muscle biopsy (in order to ensure that a sample taken would be of muscle and not just fat and fascia)
* Use of aspirin or non-steroidal anti-inflammatory agents 3 days prior to the procedure

Note: An SBMA patient who meets any of the following criteria will be excluded from the whole body MRI:

* Patient has a history of prior treatment with androgen reducing agents including LHRH agonists or antagonists, androgen receptor antagonists and selective androgen receptor modifiers.
* Patient is unable to complete the study assessments of QMT or timed walk tests.
* Patient anticipates making major lifestyle changes during the observation period relating to diet and exercise.

A Healthy Control participant who meets any of the following criteria will be excluded from the study:

* PT/PTT values that are prolonged greater than or equal to 3 seconds from the upper limit of normal (including treatment with oral and parenteral anticoagulants)
* INR greater than or equal to 1.5, thrombocytopenia (<70,000), or abnormal bleeding time or platelet dysfunction
* History of a bleeding disorder
* Use of anticoagulants

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Clinical with a confirmatory genetic testing result that is consistent with a diagnosis of spinal and bulbar muscular atrophy.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Disease progression as measured by clinical and molecular tests | Baseline to visits every 6 months to 2 years
  Clinical measurements include MRI, DEXA, physical function, swallow, and pulmonary testing. Molecular measurements include serum and plasma biomarkers, muscle analysis, and urine testing.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Grunseich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rhodes LE, Freeman BK, Auh S, Kokkinis AD, La Pean A, Chen C, Lehky TJ, Shrader JA, Levy EW, Harris-Love M, Di Prospero NA, Fischbeck KH. Clinical features of spinal and bulbar muscular atrophy. Brain. 2009 Dec;132(Pt 12):3242-51. doi: 10.1093/brain/awp258. PMID 19846582
- [Background] Atsuta N, Watanabe H, Ito M, Banno H, Suzuki K, Katsuno M, Tanaka F, Tamakoshi A, Sobue G. Natural history of spinal and bulbar muscular atrophy (SBMA): a study of 223 Japanese patients. Brain. 2006 Jun;129(Pt 6):1446-55. doi: 10.1093/brain/awl096. Epub 2006 Apr 18. PMID 16621916
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000428-N.html